CLINICAL TRIAL: NCT06600763
Title: The Effect of Ice Pack and Lukewarm Gel Pad Use on Pain, Anxiety Level and Physiological Parameters of the Child During Surgical Drain Removal in Children Aged 9-18 Years
Brief Title: Ice Pack and Lukewarm Gel Pad Use on Pain, Anxiety Level and Physiological Parameters
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Abdurrahman Başkurt, Nursing, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024/82
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Pain; Anxiety; Children; Surgery
Keywords: pain; anxiety; children; surgery
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ice pack (Experimental): Ice pack application group: An ice pack kept in the refrigerator and having a temperature of -10 degrees Celsius will be wrapped in sterile gauze and applied to the drain area of the pediatric patient who is decided to end the surgical drain indication. The temperature of the area where the ice pack is applied will be measured at one minute intervals, and when the relevant area reaches a temperature of 13.6 0C, the physician will be informed and the drain removal procedure will be initiated. The child will be asked to mark the degree of pain felt before, during and after the procedure.
  Interventions: Other: Ice pack
- warm gel (Experimental): Warm gel pad application group: Gel pads kept at room temperature will be applied to the drain area of the pediatric patient whose surgical drain indication is decided to end, in a sheath designed to wrap around the drain. After waiting for 10 minutes in the application area, the drainage system will be removed by the physician.
  Interventions: Other: warm gel pad
- Control (No Intervention): Control group: The integrated drainage system will be withdrawn by the physician. The child will not receive any non-pharmacologic intervention before, during or after the procedure.

INTERVENTIONS:
Other: Ice pack — The temperature of the area where the ice pack is applied will be measured at one minute intervals, and when the relevant area reaches a temperature of 13.6 0C, the physician will be informed and the drain removal procedure will be initiated.
  Arms: Ice pack
Other: warm gel pad — Gel pads kept at room temperature will be applied to the drain area of the pediatric patient whose surgical drain indication is decided to end, in a sheath designed to wrap around the drain. After waiting for 10 minutes in the application area, the drainage system will be removed by the physician.
  Arms: warm gel

SUMMARY:
The study was planned as a randomized controlled experimental study to determine the effect of cold application used during surgical drain removal on pain, anxiety level and physiological parameters of children aged 9-18 years.

The study will be conducted between July 2024 and April 2025 in the Pediatric Surgery Service of Adana City Training and Research Hospital. Pediatric Surgery Service has a capacity of 24 beds and 14 nurses work on a roster basis with 5 nurses during the day and 3 nurses at night. The clinical physician staff consists of 8 pediatric surgery specialists and 1 pediatric urologist. Mostly, acute abdomen, intra-abdominal mass excision, hypospadias surgery and congenital megacolon surgeries are performed.

The clinic provides outpatient and emergency services on a 24/7 basis. Data Collection In the study, children treated in pediatric surgery and followed up with drainage system after abdominal surgery will be evaluated in terms of sampling criteria and children who do not meet the criteria will be excluded from the study.

Application

1. Phase: The necessary ethics committee and institutional permission will be obtained before starting the study.
2. Stage: The decision to remove the drainage system after the end of function or end of indication is communicated to the investigator by the physician.
3. Stage: After obtaining written informed consent from the child's parents for the drain removal procedure, the researcher will explain the drain removal procedure and what will be done during the procedure to the parents. Then the descriptive information form will be filled.
4. Stage: Physiological parameters (pulse, blood pressure, respiration, SPO2 ) of the children will be measured by the researcher before and after the procedure.
5. Before the procedure, the necessary materials (ice pack or warm gel ice, infrared thermometer, gloves, saline, scalpel, clamp, sterile sponge, plaster and scissors) will be prepared and the drainage system will be clamped.
6. The parent and nurse will assess and record the child's pain score 15 minutes before, during and 15 minutes after the procedure. The child will be asked to make the same assessments and the results will be recorded.

DETAILED DESCRIPTION:
Non-pharmacologic methods can be used to reduce pain during drain removal. One of these methods is cold application. Cold application shows a local anesthetic effect in the application area by increasing the release of endogenous opioids by stimulating touch receptors based on the gate control theory and the pain felt is reduced as a result of these mechanisms.

It is thought that ice pack and warm gel ice applications to be used during drain removal in pediatric patients may be a non-pharmacologic method for surgical drain removal and will contribute to comprehensive research on this subject.

The study was planned as a randomized controlled experimental study to determine the effect of cold application used during surgical drain removal on pain, anxiety level and physiological parameters of children aged 9-18 years.

The study will be conducted between July 2024 and April 2025 in the Pediatric Surgery Service of Adana City Training and Research Hospital. Pediatric Surgery Service has a capacity of 24 beds and 14 nurses work on a roster basis with 5 nurses during the day and 3 nurses at night. The clinical physician staff consists of 8 pediatric surgery specialists and 1 pediatric urologist. Mostly, acute abdomen, intra-abdominal mass excision, hypospadias surgery and congenital megacolon surgeries are performed.

The clinic provides outpatient and emergency services on a 24/7 basis. Data Collection In the study, children treated in pediatric surgery and followed up with drainage system after abdominal surgery will be evaluated in terms of sampling criteria and children who do not meet the criteria will be excluded from the study.

Application

1. Phase: The necessary ethics committee and institutional permission will be obtained before starting the study.
2. Stage: The decision to remove the drainage system after the end of function or end of indication is communicated to the investigator by the physician.
3. Stage: After obtaining written informed consent from the child's parents for the drain removal procedure, the researcher will explain the drain removal procedure and what will be done during the procedure to the parents. Then the descriptive information form will be filled.
4. Stage: Physiological parameters (pulse, blood pressure, respiration, SPO2 ) of the children will be measured by the researcher before and after the procedure.
5. Before the procedure, the necessary materials (ice pack or warm gel ice, infrared thermometer, gloves, saline, scalpel, clamp, sterile sponge, plaster and scissors) will be prepared and the drainage system will be clamped.
6. The parent and nurse will assess and record the child pain score 15 minutes before, during and 15 minutes after the procedure. The child will be asked to make the same assessments and the results will be recorded.

Ice pack application group: An ice pack kept in the refrigerator and having a temperature of -10 degrees Celsius will be wrapped in sterile gauze and applied to the drain area of the pediatric patient who is decided to end the surgical drain indication. The temperature of the area where the ice pack is applied will be measured at one minute intervals, and when the relevant area reaches a temperature of 13.6 0C, the physician will be informed and the drain removal procedure will be initiated. The child will be asked to mark the degree of pain felt before, during and after the procedure.

Warm gel pad application group: Gel pads kept at room temperature will be applied to the drain area of the pediatric patient whose surgical drain indication is decided to end, in a sheath designed to wrap around the drain. After waiting for 10 minutes in the application area, the drainage system will be removed by the physician.

Control group: The integrated drainage system will be withdrawn by the physician. The child will not receive any non-pharmacologic intervention before, during or after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between the ages of 9 and 18,
* The child does not have developmental delay (Developmental Problems: Delay in one or more of the developmental areas such as communication, social-emotional, cognitive, sensory functions, fine-rough movements, self-care, loss of function, loss of ability, loss of ability, limitation of participation in life as a result of disease)
* Follow-up with surgical drain
* The child does not have a chronic disease that may affect his/her life
* Voluntariness of the parent and child to participate in the study

Exclusion Criteria:

* The child is under 9 years of age
* Communication problems
* Not volunteering to participate in the study
* Presence of more than one surgical drain
* The presence of developmental delay in the child (Developmental Problems: Delay in one or more of the developmental areas such as communication, social-emotional, cognitive, sensory functions, fine-rude movements, self-care, loss of function, loss of ability, loss of ability, restriction of participation in life as a result of disease)
* Previous surgical procedure under general anesthesia
* Use of any analgesic medication until at least 6 hours before the procedure

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
State-Trait Continuity Inventory for Children | 1 hour
  State-Trait Continuity Inventory for Children : The inventory, which is used to measure the state and trait anxiety states of children, was developed by Spielberger in 1973. It is a simplified form of the State-Trait Anxiety Inventory developed for adults for children. While the number of options was 4 in the adult form, it was reduced to 3 in the child form. Özusta translated the inventory into Turkish and conducted an application study.
Pain level | 1 hour
  Numerical Pain Scale : This method, which aims to determine the severity of pain, aims to explain the patient's pain in numbers. On numerical scales, absence of pain (0) is evaluated as unbearable pain (10).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Simsek Yaban Z, Alvarez-Garcia C, Bozdemir H. The effect of cold application on pain during the chest tube removal: A meta-analysis. Turk Gogus Kalp Damar Cerrahisi Derg. 2023 Jul 27;31(3):398-407. doi: 10.5606/tgkdc.dergisi.2023.23846. eCollection 2023 Jul. PMID 37664777
- [Result] Kazan AGDEE. (2011). Soğuk Uygulamalar ve Hemşirelik Bakımı. HUHEMFAD. 18(1):73-82.
- [Result] Knowlton MC. Nurse's guide to surgical drain removal. Nursing. 2015 Sep;45(9):59-61. doi: 10.1097/01.NURSE.0000470418.02063.ca. No abstract available. PMID 26287712
- [Result] Özveren, H. (2011). Ağrı kontrolünde farmakolojik olmayan yöntemler. Sağlık Bilimleri Fakültesi Hemşirelik Dergisi, 18(1), 83-92.
- [Result] Ertug N, Ulker S. The effect of cold application on pain due to chest tube removal. J Clin Nurs. 2012 Mar;21(5-6):784-90. doi: 10.1111/j.1365-2702.2011.03955.x. Epub 2011 Nov 15. PMID 22082021